CLINICAL TRIAL: NCT02375711
Title: Evaluation of Immunosenescence as a Predictive Biomarker of HBV Vaccine Efficacy in Chronic Renal Disease Patient
Brief Title: Immunosenescence and Hepatitis B Virus (HBV) Vaccine Efficacy in Chronic Renal Disease Patient
Acronym: IVVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems in including patients in the study
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2013/173
Record Dates: First submitted 2014-04-09; First posted 2015-03-03 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01

CONDITIONS: Chronic Renal Disease
Keywords: Chronic renal disease; Hepatitis B vaccine; Biological Aging
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic Renal Failure (Experimental): Patients with renal failure, with creatinine clearance between 60 and 15 ml/min. A blood sample is achieved at 0, 1, 3 and 6 months.
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — A blood sample of 35 ml is achieved at 1 month to evaluate the anti-HBV cell response. Two other blood samples of 10 ml are scheduled 3 and 6 months after vaccination to assess humoral response to HBV vaccination.

SUMMARY:
The aim of this study is to investigate the role of immunosenescence in the HBV vaccination response in patients with renal insufficiency.

DETAILED DESCRIPTION:
The risk of infection with hepatitis B during exposure to blood is high (30% against 1.8% for Hepatitis C Virus and HIV 1%) and dialysis patients are a population at risk. Vaccination against this virus, which is very effective in the general population (vaccine response: 90 to 95%), is highly recommended in dialysis patients. However, numerous studies have shown that HBV vaccination was less effective in patients with chronic renal disease than in the general population. The reasons for low vaccine response are poorly understood. However, recent data suggest that renal failure could induce accelerated immunosenescence.

The aging of the immune system, or immunosenescence, is a complex and profound phenomenon of the immune system during life. The gradual reduction of the generation of naive T cells in the thymus is the major cause of immunosenescence. But this process is also associated with an accumulation of lymphocytes at the end of differentiation.

In this context, the decrease in vaccine response and increased infections in renal insufficiency might be correlated, as in the elderly population, with the aging of the immune system. The aim of this study is to investigate the role of immunosenescence in the HBV vaccination response in patients with renal insufficiency.

Vaccination against HBV is not performed for the purposes of the study, but due to the existing vaccine indication for the subject. Included patients receive vaccination as routine care according to the recommendations and the vaccination schedule recommended by the Health Authority.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication of HBV vaccination
* Patient with renal disease, with a creatinine clearance between 15 and 60ml/min
* Patient who have never been vaccinated against HBV
* Patient with negative serology for HBV
* Patient able to understand the reason of the study
* Patient not opposed to the conservation of biological samples for scientific research

Exclusion Criteria:

* Patient infected with Hepatitis B or with history of vaccination against HBV
* Patient suffering from psychotic illness
* Patient with any history of immunosuppressive therapy
* Patient with infectious and/or cancer diseases in evolution

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Cluster of Differentiation (CD) 8+ CD 57+ CD 28- / CD 8+ T lymphocytes Ratio in Peripheral Blood | 13 months
  The primary outcome is assessed 1 month after the vaccination schedule. The percentage of CD 8+ and CD 8+ CD 28- CD 57+ lymphocytes were determined by flow cytometry.

SECONDARY OUTCOMES:
Calculated Creatinine Clearance (Cockcroft-Gault Equation) | 13 months
  Creatinine clearance calculated using Cockcroft-Gault equation and adjusted for body surface area. Calculated Creatinine Clearance: method to approximate kidney function. It measures rate creatinine (substance formed from metabolism of creatine) is cleared from blood by kidneys.
Interferon gamma and Interleukin-10 production of Peripheral blood T lymphocytes | 13 months
  Analysis of cytokine production is assessed by flow cytometry after stimulation of lymphocytes T.
Percentage of Lymphocytes subpopulations in Peripheral Blood Mononuclear Cells | 13 months
  Different lymphocyte subpopulations will be quantified by flow cytometry using the following antibodies: CD 3, CD 4, CD 8, CD 19, CD 25, CD 27, CD 28, CD 31, CD 45RO, CD 45RA, CD 56, CD 62L, Cytotoxic T-Lymphocyte Antigen 4, Programmed cell death protein 1, CD 38, CD 127, Forkhead box P3.
T-cell receptor excision circle (TREC) level in peripheral blood mononuclear cells (PBMC) | 13 months
  TREC study used a technique of quantitative Polymerase Chain Reaction performed on DNA extracted from PBMC.

OTHER OUTCOMES:
Body Mass Index | at patient inclusion
  body mass index= body weight (kg) divided by square of body height (m2)
Cytomegalovirus (CMV) serology | 18 months
  Modeling of vaccine efficacy using a multivariate logistic regression will investigate whether there is a link between immunosenescence and vaccine response, adjusting on factors influencing the immunosenescence as CMV status.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile COURIVAUD, Doctor, Principal Investigator — University Hospital, Inserm UMR 1098, Besançon
Locations (1):
- Service de néphrologie, CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No